CLINICAL TRIAL: NCT07280234
Title: Comparison of Intradermal Microinjections of Tanexamic Acid and Oral Tranexamic Acid in the Management of Melasma. A Randomized Controlled Trial.
Brief Title: Comparison of Intradermal Microinjections of Tanexamic Acid and Oral Tranexamic Acid in the Management of Melasma.
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Hayat Abad Medical Complex, Peshawar (Other Government)
Responsible Party: Principal Investigator, Syeda Sana Zaman, Trainee Medical Officer, Hayat Abad Medical Complex, Peshawar
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HayatabadHMC
Record Dates: First submitted 2025-11-28; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Melasma
Keywords: Melasma
MeSH Terms: conditions — Melanosis | interventions — Tranexamic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intradermal microinjections of Tranexamic Acid (Active Comparator): In this group patients will recieve intradermal microinjections of tranexamic acid
  Interventions: Drug: Intradermal microinjections of tranexamic acid
- Oral tranexamic acid (Active Comparator): In this group patients will recieve oral tranexamic acid
  Interventions: Drug: Oral tranexamic acid

INTERVENTIONS:
Drug: Intradermal microinjections of tranexamic acid — This group A will recieve intradermal microinjections of tranexamic acid
  Arms: Intradermal microinjections of Tranexamic Acid
Drug: Oral tranexamic acid — This group B will recieve oral tranexamic acid
  Arms: Oral tranexamic acid

SUMMARY:
In this study we compared the effect of intradermal microinjections of tranexamic acid vs oral tranexamic acid in treatment of melasma. Given the high prevalence of melasma in Pakistan and the significant psychosocial impact on patients, particularly in Peshawar, this study will provide valuable insights into optimal treatment strategies

DETAILED DESCRIPTION:
Melasma appears as clearly established, symmetrically organised lighter patches that primarily develop on face areas that are exposed to sunlight. 1, 2 The mechanisms behind melasma remain poorly understood; nevertheless, it has been determined that this disorder becomes far more common among women of darker skin tones. 3, 4 Hormonal factors involving oral contraceptives, chronic skin inflammation, pregnancy and extended exposure to sunlight significantly impact etiopathogenesis as well as progression of melasma. 5,6 Furthermore, melasma demonstrates a higher prevalence among females, with studies suggesting that women are 9-10 times more predisposed to this disorder as compare to men.7 The occurrence of melasma within women during their pregnancy is considerably elevated, reaching as high as 63% . Pregnancy is a prevalent contributory factor to melasma whereas for men, the leading risk factors is sun exposure as well as relatives with a history of condition.7 Topical sunscreens are crucial in treatment of melasma, which should be tailored to achieve optimal effectiveness for controlling pigmentary disorders.8 However, it is typical for patients to apply 50% of suggested dosage of sunscreens on skin. Therefore, it is suggested for people with pigmentary conditions to use products that have greater SPF values. 9 Tranexamic acid (TXA) is a compound that comes from amino acid lysine. Hypopigmentation influence arises from its antiplasmin operation, which displays a structural analogy to tyrosine.5 The administration of oral TXA results in notable reduction in mMASI scores among patients of melasma.10 The administration of TXA via intradermal injection illustrates efficacy in managing both dermal as well as mixed variations of melasma. TXA is a reliable and usually well-accepted medication when administered at standard dosage.11 Several approaches of administration such as topical, oral, intradermal injections, and micro-needling along with different formulations of TXA, have shown promising outcomes in the management of melasma.12 Melasma is a acquired hyperpigmentation complaint that significantly influences quality of life predominantly among female of reproductive age. TXA has emerged as an effective treatment option due to the ability to inhibit melanogenesis by blocking the interaction in melanocytes and keratinocytes. Despite individual studies supporting both routes of administration however the direct comparative data remain limited. Therefore, this study aims to compare the efficacy and safety of intradermal microinjections versus oral administration of TXA in treatment of melasma which will evidence-based guidance for optimized management strategies.

METHODOLOGY:

The methodology of this study was designed as a prospective randomized controlled trial, which was conducted in the department of dermatology at Lady Reading Hospital from 15-November-2024 to 15-May-2025, after acquiring ethical approval from the hospital. to evaluate the comparative efficacy of intradermal tranexamic acid microinjections (TXA ID) versus oral tranexamic acid (TXA Oral) in management of melasma. The study was carried out at a tertiary care dermatology center over a period of 12 months with ethical approval obtained from the institutional review board prior to commencement. Written informed consent was secured from all subjects after a detailed explanation of study protocol potential benefits and possible side effects.

Written informed consent was acquired from all participants We enrolled 218 patients, using the previous mMASI score of intradermal tranexamic acid microinjections (TXA ID) 7.62±1.64 and 8.3±1.9213 of TXA Oral, with power 80% and confidence interval 95%. Patients aged 18 to 55 years, with clinically confirmed melasma of at least 6 months duration, Fitzpatrick skin types III-V and no active dermatological conditions in the treatment area. Exclusion criteria encompassed pregnancy or lactation, history of thromboembolic disorders, use of hormonal therapies or photosensitizing medications, recent melasma treatments within the past 3 months and known hypersensitivity to tranexamic acid. Baseline assessments included detailed medical history clinical examination and standardized digital photography under controlled lighting.

Patients were randomly allocated into two treatment groups using blocked randomization. Group A comprising 109 patients received intradermal microinjections of tranexamic acid (4 mg/ml) administered weekly using a 30-gauge insulin syringe. The injections were delivered in the affected facial areas with approximately 0.05 ml per injection point spaced 1 cm apart. Group B also consisting of 109 patients was prescribed TXA Oral at a dose of 250 mg twice daily. Both groups were instructed to use a broad-spectrum sunscreen with SPF 50 throughout the study period and were advised to maintain their usual photoprotection measures.

The primary outcome measure was the change in modified Melasma Area and Severity Index (mMASI) scores from baseline to week 8 assessed by the researcher under the direction supervision of a consultant dermatologist with experience of five years or more. The treatment response was assessed using the aforementioned index as Poor response (< 25%), mild response (25 to 50%), moderate response (51 to 75%) and excellent response (> 75%). Follow-up visit was scheduled at 8-week interval for clinical evaluation, mMASI scoring and monitoring of treatment adherence.

SPSS 26 was used for analyzing the data. Age, duration of melasma, pre and post treatment mMASI scores were expressed as mean ± standard deviation while gender and clinical profile were presented as frequencies and percentages. Paired t-tests were used to compare pre- and post-treatment mMASI scores within groups, while independent t-tests assessed differences between groups. Chi-square tests evaluated treatment response, with p-values <0.05 considered statistically notable.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 to 55 years, with clinically confirmed melasma of at least 6 months duration.
2. Fitzpatrick skin types III-V and no active dermatological conditions in the treatment area.

Exclusion Criteria:

1. pregnancy or lactation
2. History of thromboembolic disorders
3. Use of hormonal therapies or photosensitizing medications
4. Recent melasma treatments within the past 3 months
5. Known hypersensitivity to tranexamic acid.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 218 (Actual)
Dates: Start 2024-11-14 (Actual); Primary Completion 2025-05-15 (Actual); Study Completion 2025-05-15 (Actual)

PRIMARY OUTCOMES:
Assessment of Melasma Area and Severity Index | Six months
  The primary outcome measure was the change in modified Melasma Area and Severity Index (mMASI) scores from baseline to week 8 assessed by the researcher under the direction supervision of a consultant dermatologist with experience of five years or more. The treatment response was assessed using the aforementioned index as Poor response (< 25%), mild response (25 to 50%), moderate response (51 to 75%) and excellent response (> 75%). Follow-up visit was scheduled at 8-week interval for clinical evaluation, mMASI scoring and monitoring of treatment adherence.

CONTACTS AND LOCATIONS:
Overall Officials: Ghafoor Ullah Ullah, FCPS part 2, Principal Investigator — MTI-HMC Peshawar, Peshawar Khyber PakhtunKhwa 25000
Locations (1):
- MTI-HMC Peshawar, Peshawar Khyber Pakhtunkhwa, Peshawar, Khyber Pakhtunkhwa, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided